CLINICAL TRIAL: NCT02550470
Title: Evaluation of Micropore's SpiraLith TM Absorbents Into Anesthesia Breathing Circuits
Brief Title: Evaluation of Micropore"s SpiraLith Absorbents
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Jean Daniel Eloy, MD, Assistant Professor, Department of Anesthsiology, NJMS, Rutgers, The State University of New Jersey
Other Study IDs: PRO20140001012
Record Dates: First submitted 2015-09-03; First posted 2015-09-15 (Estimated); Results first posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-02

CONDITIONS: Airway Management During Operative Procedure
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Randomized to Micropore SpiraLith: lithium hydroxide was studied for use in anesthesia as a possible replacement for calcium absorbents. This agent has been used for CO2 absorption in the military and in aerospace for over 50 years due to its high capacity and efficiency in the removal of CO2. It was however not considered usable by the medical industry due to concerns with its granular form. It has now been demonstrated that LiOH does not interact with commonly used inhalation anesthetic agents and appears to have higher CO2 removal capability.7,8
  Interventions: Device: Micropore SpiraLith; Drug: Sevoflurane
- Randomized to Drager 800 Absorbent: Calcium hydroxide lime is one of the newer clinically available carbon dioxide absorbents and probably considered the current standard of care. It is mainly composed of calcium hydroxide and calcium chloride and contains two setting agents: calcium sulfate and polyvinylpyrrolidine which contribute to the increased hardness and porosity of this absorbent. The most significant advantage of calcium hydroxide lime over other agents is that it is produced without sodium and potassium hydroxide which are strong bases.
  Interventions: Device: Carbon Dioxide Absorbents; Drug: Sevoflurane
- Randomized to Drager Free: Calcium hydroxide lime is one of the newer clinically available carbon dioxide absorbents and probably considered the current standard of care. It is mainly composed of calcium hydroxide and calcium chloride and contains two setting agents: calcium sulfate and polyvinylpyrrolidine which contribute to the increased hardness and porosity of this absorbent. The most significant advantage of calcium hydroxide lime over other agents is that it is produced without sodium and potassium hydroxide which are strong bases.
  Interventions: Device: Carbon Dioxide Absorbents; Drug: Sevoflurane

INTERVENTIONS:
Device: Carbon Dioxide Absorbents — Calcium hydroxide lime is one of the newer clinically available carbon dioxide absorbents and probably considered the current standard of care. It is mainly composed of calcium hydroxide and calcium chloride and contains two setting agents: calcium sulfate and polyvinylpyrrolidine which contribute to the increased hardness and porosity of this absorbent. The most significant advantage of calcium hydroxide lime over other agents is that it is produced without sodium and potassium hydroxide which are strong bases.
  Groups: Randomized to Drager 800 Absorbent; Randomized to Drager Free
Device: Micropore SpiraLith — lithium hydroxide was studied for use in anesthesia as a possible replacement for calcium absorbents. This agent has been used for CO2 absorption in the military and in aerospace for over 50 years due to its high capacity and efficiency in the removal of CO2. It was however not considered usable by the medical industry due to concerns with its granular form. It has now been demonstrated that LiOH does not interact with commonly used inhalation anesthetic agents and appears to have higher CO2 removal capability.
  Groups: Randomized to Micropore SpiraLith
Drug: Sevoflurane

SUMMARY:
This is an observational study investigating the duration of use and cost of the new CO2 absorbent Micropore's Spiralith®, compared to Drägersorb® 800+, Drägersorb® Free.

DETAILED DESCRIPTION:
The Principal Investigator will obtain IRB approval under expedited review. No patient written informed consent will be required as this is a process improvement minimal risk study that does not necessitates use of patient Protected Health Information. Participants will not be actually enrolled. There will be no change to the standard of care resulting from data collection on CO2 absorbent use, and no patient identifiers will be exposed. The study will take place in three operating rooms, three rooms equipped with Drager Appollo® anesthesia workstations (Draeger Medical Inc., USA) requiring use of CLIC style absorbents. An unblinded member of the research team will have access to the randomization schedule and will be responsible to place Drägersorb® 800+, Drägersorb® Free, or Micropore SpiralithTM absorbents in the designated operating rooms with three Appollo® (CLIC style absorbent). The randomly selected absorbent will be loaded on the anesthesia workstation prior to the patient's arrival in the operating room and the date, time and randomization coding will be marked on the cassette as it appears on the randomization schedule. The anesthesia providers will use low flow anesthesia with or without Sevoflurane in the 3 selected operating rooms. The practice at this institution is to use a semi-closed breathing circuit and maintain a fresh gas flow rate of approximately 2L/min with a selected tidal volume of 6-8 mL/Kg during the maintenance phase of the procedure. Flow rate would be approximately 10 L/min during the induction of anesthesia. The investigators will document time that is required to achieve 90% of the sevoflurane target concentration. These guidelines will be clearly indicated on the anesthesia workstation to ensure consistency across the multiple providers. Data logger files will be saved at the end of each case using the same coding label as the marked cassette. When the absorbent is replaced, the date and time of removal should be clearly marked on the cassette. This same date and time information should also be recorded on the source document ensuring that operating room numbers and anesthesia workstations are clearly and accurately recorded. In order to maintain the anesthesia provider blinded to the type of absorbent used, a white sheet of paper will be taped around the outside of the cassette compartment. The time that the patient is connected and disconnected from the breathing circuit must be recorded on the source document. In addition the investigators will document The absorbent unit will be replaced when the inspiratory CO2 concentration (obtained from the inspiratory limb of the breathing circuit) reaches 4 mmHg. This is an acceptable maximal inspiratory CO2 concentration which leaves sufficient time to complete a case, thereby avoiding cassette replacement during anesthesia. The anesthesia workstation fresh gas flows will be turned off at the time that the patient is disconnected from the breathing circuit to avoid variability in absorbent water content.

The absorbing capacity of the cassettes will be determined by calculating the duration of absorbent use from the time of first use to the time of cassette removal. Each absorbent will be evaluated through a total of 5 rounds. We expect to have about 60 surgeries for each absorbent. Averaged duration of absorbent use will be compared between different types of absorbents (Drägersorb® 800+, Drägersorb® Free, Micropore SpiralithTM).

ELIGIBILITY:
Inclusion Criteria:

* All comers to the 3 designated Operating Rooms.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients scheduled for surgery in the selected OR Rooms
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2015-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J.Daniel Eloy, MD, Principal Investigator — Rutgers University
Locations (1):
- University Hospital, Newark, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were not actually enrolled. The randomly selected absorbent was loaded on the anesthesia workstation prior to the patient's arrival in the operating room.
Pre-assignment Details: The number of participants is unknown as participants were not enrolled. The Enrollment number in the Protocol section is reporting the number of surgeries.
Units Other Than Participants: Absorbent units
Groups:
- Randomized to Micropore SpiraLith: lithium hydroxide was studied for use in anesthesia as a possible replacement for calcium absorbents. This agent has been used for CO2 absorption in the military and in aerospace for over 50 years due to its high capacity and efficiency in the removal of CO2. It was however not considered usable by the medical industry due to concerns with its granular form. It has now been demonstrated that LiOH does not interact with commonly used inhalation anesthetic agents and appears to have higher CO2 removal capability.7,8
  Micropore SpiraLith: lithium hydroxide was studied for use in anesthesia as a possible replacement for calcium absorbents. This agent has been used for CO2 absorption in the military and in aerospace for over 50 years due to its high capacity and efficiency in the removal of CO2. It was however not considered usable by the medical industry due to concerns with its granular form. It has now been demonstrated that LiOH does not interact with commonly used inhalation anesthetic agents and appears to have higher CO2 removal capability.
  Sevoflurane
- Randomized to Drager 800 Absorbent; Randomized to Drager Free: Calcium hydroxide lime is one of the newer clinically available carbon dioxide absorbents and probably considered the current standard of care. It is mainly composed of calcium hydroxide and calcium chloride and contains two setting agents: calcium sulfate and polyvinylpyrrolidine which contribute to the increased hardness and porosity of this absorbent. The most significant advantage of calcium hydroxide lime over other agents is that it is produced without sodium and potassium hydroxide which are strong bases.
  Carbon Dioxide Absorbents: Calcium hydroxide lime is one of the newer clinically available carbon dioxide absorbents and probably considered the current standard of care. It is mainly composed of calcium hydroxide and calcium chloride and contains two setting agents: calcium sulfate and polyvinylpyrrolidine which contribute to the increased hardness and porosity of this absorbent. The most significant advantage of calcium hydroxide lime over other agents is that it is produced without sodium and potassium hydroxide which are strong bases.
  Sevoflurane
Period: Overall Study
Arm/Group | Randomized to Micropore SpiraLith | Randomized to Drager 800 Absorbent | Randomized to Drager Free
Started | NA; 58 Absorbent units (time to reach FiO2 of 4 mm Hg was recorded for each absorbent in the anesthesia circuit Absorbent units other than participants were assigned to Arms/Groups) | NA; 65 Absorbent units (time to reach FiO2 of 4 mm Hg was recorded for each absorbent in the anesthesia circuit Absorbent units other than participants were assigned to Arms/Groups) | NA; 63 Absorbent units (time to reach FiO2 of 4 mm Hg was recorded for each absorbent in the anesthesia circuit Absorbent units other than participants were assigned to Arms/Groups)
Completed | NA; 58 Absorbent units (time to reach FiO2 of 4 mm Hg was recorded for each absorbent in the anesthesia circuit Absorbent units other than participants were assigned to Arms/Groups) | NA; 65 Absorbent units (time to reach FiO2 of 4 mm Hg was recorded for each absorbent in the anesthesia circuit Absorbent units other than participants were assigned to Arms/Groups) | NA; 63 Absorbent units (time to reach FiO2 of 4 mm Hg was recorded for each absorbent in the anesthesia circuit Absorbent units other than participants were assigned to Arms/Groups)
Not Completed | NA; 0 Absorbent units | NA; 0 Absorbent units | NA; 0 Absorbent units

BASELINE CHARACTERISTICS:
Population: Absorbent units other than participants were assigned to Arms/Groups
Units Other Than Participants: Absorbent units
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized to Micropore SpiraLith | Randomized to Drager 800 Absorbent | Randomized to Drager Free | Total
Number analyzed (Participants) | NA | NA | NA | NA
Number analyzed (Absorbent units) | 58 | 65 | 63 | 186
Age, Categorical [Count of Units; unit: Absorbent units] — The randomly selected absorbent were loaded on the anesthesia workstation prior to the patient's arrival at the operating room. Patients of any age were not actually enrolled.
  Absorbent units
    <=18 years | NA — The randomly selected absorbent was loaded on the anesthesia workstation prior to the patient's arrival at the operating room. Patients were not actually enrolled | NA — The randomly selected absorbent was loaded on the anesthesia workstation prior to the patient's arrival at the operating room. Patients were not actually enrolled | NA — The randomly selected absorbent was loaded on the anesthesia workstation prior to the patient's arrival at the operating room. Patients were not actually enrolled | NA — Total not calculated because data are not available (NA) in one or more arms.
    Between 18 and 65 years | NA — The randomly selected absorbent was loaded on the anesthesia workstation prior to the patient's arrival at the operating room. Patients were not actually enrolled | NA — The randomly selected absorbent was loaded on the anesthesia workstation prior to the patient's arrival at the operating room. Patients were not actually enrolled | NA — The randomly selected absorbent was loaded on the anesthesia workstation prior to the patient's arrival at the operating room. Patients were not actually enrolled | NA — Total not calculated because data are not available (NA) in one or more arms.
    >=65 years | NA — The randomly selected absorbent was loaded on the anesthesia workstation prior to the patient's arrival at the operating room. Patients were not actually enrolled | NA — The randomly selected absorbent was loaded on the anesthesia workstation prior to the patient's arrival at the operating room. Patients were not actually enrolled | NA — The randomly selected absorbent was loaded on the anesthesia workstation prior to the patient's arrival at the operating room. Patients were not actually enrolled | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Units; unit: Absorbent units] — The randomly selected absorbent was loaded on the anesthesia workstation prior to the patient's arrival at the operating room. Patients were not actually enrolled
  Absorbent units
    Female | NA — The randomly selected absorbent was loaded on the anesthesia workstation prior to the patient's arrival at the operating room. Patients were not actually enrolled | NA — The randomly selected absorbent was loaded on the anesthesia workstation prior to the patient's arrival at the operating room. Patients were not actually enrolled | NA — The randomly selected absorbent was loaded on the anesthesia workstation prior to the patient's arrival at the operating room. Patients were not actually enrolled | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | NA — The randomly selected absorbent was loaded on the anesthesia workstation prior to the patient's arrival at the operating room. Patients were not actually enrolled | NA — The randomly selected absorbent was loaded on the anesthesia workstation prior to the patient's arrival at the operating room. Patients were not actually enrolled | NA — The randomly selected absorbent was loaded on the anesthesia workstation prior to the patient's arrival at the operating room. Patients were not actually enrolled | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Duration of Use Under Clinical Anesthesia of Each Absorbent
Description: Average lifespan of Spiralith® (minutes), Drägersorb® 800 Plus (minutes), Drägersorb® Free (minutes)
Time Frame: Assesed for the duration of each absorbent's use, up to 5 days
Population: Patients were not actually enrolled. Overall number of surgeries are provided
Measure: Mean (Standard Deviation); unit: min
Units Other Than Participants: Absorbent units
Arm/Group | Randomized to Micropore SpiraLith | Randomized to Drager 800 Absorbent | Randomized to Drager Free
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Absorbent units) | 58 | 65 | 63
min | 1931 (472) | 1806 (343) | 1527 (295)

2. Secondary Outcome: Cost of Each Absorbent's Use
Time Frame: Assesed for the duration of each absorbent's use, up to 5 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: At Risk represents surgeries, number of participants unknown as participants were not enrolled
Arm/Group | Randomized to Micropore SpiraLith | Randomized to Drager 800 Absorbent | Randomized to Drager Free
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/65 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/65 | 0/63
Other Adverse Events (participants affected / at risk) | 0/58 | 0/65 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No